CLINICAL TRIAL: NCT07385937
Title: Effectiveness of Genistein on the Progression of Cognitive Impairment in Patients With Mild Cognitive Impairment: Controlled Clinical Trial
Brief Title: Effectiveness of Genistein in Mild Cognitive Impairment
Acronym: EXTRAGENIAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UCAMCFE-00040
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease (AD); Mild Cognitive Impairment (MCI)
Keywords: Genistein; Dementia; Cognitive impairment; Neuroprotection; Prevention
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia | interventions — Genistein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The product will have the same characteristics as the experimental product.
  Interventions: Dietary Supplement: Control product placebo
- Genistein (Experimental): Subjects will consume two capsules daily. Each capsule will be taken before the two main meals, each 100 mg tablet.
  Interventions: Dietary Supplement: Genistein

INTERVENTIONS:
Dietary Supplement: Genistein — Soy isoflavone
  Arms: Genistein
Dietary Supplement: Control product placebo — It will be supplied in a color and shape similar to the active product, but with maltodextrin, an inert substance.
  Arms: Placebo

SUMMARY:
Randomized, placebo-controlled, double-blind, multicenter clinical trial with two parallel study arms (experimental and placebo) to assess the efficacy of genistein extract consumption over 18 months on cognitive decline in patients with prodromal Alzheimer's disease.

DETAILED DESCRIPTION:
The study aims to evaluate the effect of genistein over 18 months compared to placebo on the progression of cognitive impairment in subjects diagnosed with mild cognitive impairment (MCI) due to Alzheimer's disease (AD) in the following areas:

1. Global assessment of dementia: overall evaluation of functionality and cognitive decline in MCI subjects.
2. Global cognitive functions: assessment of general cognitive abilities.
3. Episodic memory: evaluation of memory performance.
4. Activities of daily living: assessment of the ability to perform basic and instrumental daily activities.
5. Emotional and depressive state: evaluation of subjects' mood and depressive symptoms

ELIGIBILITY:
Inclusion Criteria:

* Patient over 50 years of age.
* Patient diagnosed with mild cognitive impairment (MCI) for Alzheimer's disease (AD) according to the National Institute on Aging and Alzheimer's Association (NIA-AA, 2024) criteria:

  * MMSE scores between 22 and 30 (inclusive; exceptions may be made for subjects with less than 5 years of education).
  * Evidence of concern about change in cognition, compared to the person's previous level (subjective memory complaint/impairment for more than 6 months in the past year and/or confirmed by the informant and/or physician).
  * A Clinical Dementia Rating (CDR) score of 0.5 with a memory domain score of 0.5.
  * Essentially preserved activities of daily living.
* Evidence of elevated cortical amyloid by positron emission tomography (PET) with F18-flutemetamol. • Patients will be treated pharmaceutically according to the guidelines.

Exclusion Criteria:

* Diagnosis of a significant neurological disease other than Alzheimer's disease.
* Moderate depression as assessed by a Geriatric Depression Scale (GDS-D) score >8, or any other serious psychiatric disorder.
* Taking supplements containing isoflavones.
* Having a hormone-dependent neoplastic disease.
* Diagnosis of significant cerebrovascular disease.
* Having a serious systemic illness that would prevent completion of the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The change in overall cognitive function and the deterioration in the ability to perform activities of daily living | From baseline to month 18
  The primary variable to be evaluated is the change in overall cognitive function and the deterioration in the ability to perform activities of daily living, assessed through the mean change by the Integrated Alzheimer's Disease Rating Scale (iADRS) score.
  iADRS is an assessment tool designed to comprehensively measure cognitive and functional decline in patients with Alzheimer's disease, especially in the early stages. It combines elements of cognitive and functional assessment in a single scale, using ADAS-Cog and ADCS-ADL. In this case, version ADAS-Cog14 was used.

SECONDARY OUTCOMES:
Detection and assessment of cognitive impairment | 18 months
  The Mini-Mental State Examination (MMSE) is one of the most widely used tools for detecting and assessing cognitive impairment, including Alzheimer's disease. It is a brief and simple test that evaluates various cognitive functions: spatial and temporal orientation, immediate memory, attention and calculation, delayed memory, language, praxis (naming, repetition, comprehension of verbal commands, reading, spontaneous writing and copying drawings) and visual construction.
Assess symptoms of depression | 18 months
  The GDS-15 (Geriatric Depression Scale - 15 items). This instrument was specifically designed for use in elderly populations to detect possible depression. It consists of 15 items with dichotomous yes/no responses.
Severity of dementia | 18 months
  CDR-SB: A semi-structured interview with the primary informant and the patient, evaluated according to the evaluator's clinical judgment. It assesses the domains of Memory, Orientation, Judgment and Problem Solving, Community Affairs, Home and Hobbies, and Personal Care, with greater emphasis on the first domain.
global cognition | 18 months
  ADAS-Cog: This test aims to measure the severity of dementia (global cognition, memory, language, etc.). The ADAS-Cog14 was chosen, which adds additional items (delayed word recall, digit cancellation, and maze or verbal fluency test) to the original test, improving the scale's sensitivity without significantly increasing assessment time.
Assess functionality in patients with cognitive impairment | 18 months
  The ADCS-ADL and ADCS-ADL-MCI questionnaires assess functionality but they are aimed at different populations. ADCS-ADL aims to assess functionality in activities of daily living. ADCS-ADL-MCI, on the other hand, aims to assess the impact of Mild Cognitive Impairment (MCI) on Activities of Daily Living (ADLs).
Activities of daily living | 18 months
  DAD-E: It aims to evaluate the functional impact of dementia on activities of daily living, through a questionnaire applied to the main informant.
Assess verbal memory | 18 months
  The TAVEC (Test de Aprendizaje Verbal España-Complutense) is a neuropsychological tool widely used in Spain and other Spanish-speaking countries. It aims to assess episodic verbal memory, including learning, immediate recall, delayed recall, recognition, attention, and sensitivity to interference.
Assess cognitive functions | 18 months
  The Trail Making Test (TMT) is a widely used neuropsychological test. It aims to assess processing speed, sustained and divided visual attention, visual tracking, executive functions (cognitive flexibility), and cognitive flexibility.
visuospatial abilities and visual memory | 18 months
  The Clock Drawing Test (CDT) aims to evaluate visuospatial abilities and skills, visual memory and executive functions (strategy, organization).
Assess visual memory, visuospatial perception, and executive functions | 18 months
  The Rey-Osterrieth Test is a widely used neuropsychological test for assessing visual memory, visuospatial perception, and executive functions. These functions are often affected in Alzheimer's disease, making this test useful in its assessment.
Working memory and attention | 18 months
  Digit Span: It aims to assess short-term verbal memory (forward span) and auditory-verbal working memory (reverse span), as well as attention, sequencing, and mental manipulation of information.
Ability to generate words within a specific category | 18 months
  Semantic fluency is a neuropsychological test. It aims to evaluate lexical-semantic access capacity, knowledge organization in memory, executive functions (planning, initiation, flexibility, response control), and semantic memory. This test is particularly useful for assessing executive function and language, two areas that are often affected in Alzheimer's disease.
Assess executive functions | 18 months
  The F.A.B. (Frontal Assessment Battery) is a brief neuropsychological tool designed to assess executive functions, which are often affected in Alzheimer's disease and other dementias. It aims to evaluate executive functions (conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, autonomy) by combining verbal instructions with tasks that require verbal responses or motor actions.
Knowing the amount of ß-amyloid (βA) plaques | 18 months
  Positron emission tomography is a molecular imaging technique that measures the activity of a radiopharmaceutical that marks ß-amyloid (βA) plaques through the SUV (standard uptake value), which should be based on the amount of AB and can be relativized to match the change we expect to see. The mean change from baseline to month 18 in the standard uptake value (SUV) of composite cortical amyloid will be evaluated using the amyloid tracer [18F] flutemetamol by positron emission tomography (PET) imaging.
Knowing the response to treatment | 18 months
  The inclusion of serum biomarkers may offer a more comprehensive perspective on the underlying mechanisms and response to treatment.
Comorbidities and Medication | 18 months
  Take into account associated diseases, such as hypertension, diabetes, dyslipidemia, and other chronic diseases suffered by the patient, as well as concomitant medication. Document all medications that participants are taking at the start of the study or during its course, especially those that may influence cognitive function.
Demographic variables | 18 months
  Age and gender; educational level; age and year of birth; tobacco and/or alcohol consumption.
Safety | 18 months
  The safety of investigational products (IPs) will be assessed by recording adverse events (AEs) throughout the study, i.e., from the baseline visit to the final visit and a blood test.

CONTACTS AND LOCATIONS:
Locations (1):
- UCAM HiTech, Sport & Health Innovation Hub, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No